CLINICAL TRIAL: NCT03449914
Title: Prognostic Value of Baseline G8 Geriatric Assessment in Elderly Metastatic Colorectal Cancer Patients
Brief Title: The GOLD Study: G8 in OLDer Patients
Acronym: GOLD
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Istituto Oncologico Veneto IRCCS (Other)
Collaborators: Roche Pharma AG (Industry)
Responsible Party: Sponsor
Other Study IDs: GOLD
Record Dates: First submitted 2018-02-23; First posted 2018-02-28 (Actual); Last update posted 2023-11-29 (Actual); Status verified 2023-11

CONDITIONS: Elderly Metastatic Colorectal Cancer Patients
Keywords: ECOG PS; Timed Up and Go test; G8 score

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Management of older cancer patients is challenging, due to a lack of good quality evidence to guide treatment decisions, as well as the wide variability in the level of fitness for treatment of elderly patients. Oncologists are faced with the challenge of determining the most suitable treatment for an individual taking into account their comorbidities, competing causes of death, quality of life and functional reserve.

Colorectal cancer (CRC) is the second leading cause of cancer-related deaths in the western world and ranks second among the most frequent malignancies in Europe in both men and women. The incidence and mortality of CRC strongly increases with age. Approximately 60% of new cases of CRC and 70% of CRC-related deaths occur in patients aged 65 years and older, with about 40% of patients aged 75 years or older.

The oncologists' therapeutic decision-making for elderly patients with metastatic colorectal cancer (mCRC) has been largely debated in the last few years, mainly because of the lack of trial-based recommendations, due to the underrepresentation of patients more than 65 years old in clinical trials. As a consequence, therapeutic choices in this setting are frequently driven by data from retrospective, pooled and meta-analyses. These results do not necessarily reflect the general population affected with mCRC and are often limited by potential confounding factors.

It is well recognized that chronological age is not an effective criterion on which to base therapeutic decisions. Rather, treatment tolerability in an older cancer patient is primarily related to physiological or biological age, that is the level of fitness, which takes into account factors such as functional status and comorbidities. Physiological age is better assessed with a comprehensive geriatric assessment (CGA), a multidisciplinary evaluation covering domains such as cognitive and mood status, functionality, comorbidities, and nutrition. These deficits are prevalent in older patients but which may be missed with routine evaluation.

There is now strong evidence that use of a CGA assessment in a general geriatric patient population can improve health outcomes. While some form of geriatric assessment have been recommended by specialist advisory panels for all elderly patients in whom chemotherapy is considered, evidence of CGA leading to improved outcomes in a geriatric population with cancer is very limited. CGA for older patients with cancer does appear to provide information relating to prognosis, likelihood of toxicity from chemotherapy, and has been shown to influence treatment decisions. However, this approach is time-consuming, leading cancer specialists to seek an easier screening tool that can separate fit older patients with cancer, who are able to receive standard cancer treatment, from vulnerable patients that should subsequently receive a full assessment to guide tailoring of their treatment regimen.

The G8 is a simple 8-items screening tool, developed specifically for older patients with cancer. This tool, addressed by the clinician, covers multiple domains, focusing on nutritional status, mobility, neuropsychological problems, medication use, self-rated health status and age. The G8 demonstrated a good sensitivity in identifying patients with impairments across multiple domains when a cut-off of 14 points is adopted. Patients with a score < 14 would be candidate to a CGA. Nevertheless, this cut-off showed poor specificity and negative predictive value. Furthermore, some evidences suggested that the G8 might be able to predict survival, while its predictive value for treatment-related toxicities has not been extensively explored.

While literature data support a promising role for G8 as a simple cost-effective screening tool in elderly patients, to date its use in clinical practice is not widespread, and only selected centers with a focus in geriatric oncology routinely perform this assessment to enhance the baseline evaluation of patients before treatment choice.

The lack of ''real life population'' data makes it difficult to evaluate the role of G8 in the setting of common practice in an unselected population and to prove its efficacy and reliability outside selected cases.

Moreover, recent data suggest how a physical performance test, such as Timed Up and Go, could be a useful indicators of prognosis, functional decline and treatment-related complications.

This study is designed to promote a comprehensive evaluation of elderly patients before treatment decisions and to prospectively evaluate the association of G8 assessment with clinical outcome and treatment-related severe toxicity in the real life population of elderly patients with colorectal cancer in Veneto. Additionally, preliminary data on feasibility and reliability of Timed Up and Go measurement as prognostic determinant and dynamic marker, will be collected.

ELIGIBILITY:
Inclusion Criteria:

* New diagnosis of metastatic colorectal cancer, untreated in the metastatic setting
* Age ≥ 70 years
* Availability of clinical data
* Before patient registration, written informed consent must be given according to ICH/GCP, and national/local regulations

Min Age: 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: Elderly (> 70 years) patients with metastatic colorectal cancer
Sampling Method: Non-Probability Sample
Enrollment: 109 (Actual)
Dates: Start 2017-10-26 (Actual); Primary Completion 2022-02-07 (Actual); Study Completion 2024-07 (Estimated)

PRIMARY OUTCOMES:
Evaluate the prognostic value of baseline G8 screening tool for survival. | Up to 12 months

CONTACTS AND LOCATIONS:
Locations (1):
- Istituto Oncologico Veneto IRCCS, Padua, Italy